CLINICAL TRIAL: NCT00780572
Title: Implementation of Real-Time ADE Surveillance and Decision Support
Acronym: VA ADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IAB 05-224
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Adverse Drug Events
Keywords: Safety Management; Risk Management; surveillance; triggers
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: ADE Alerts (Experimental): Arm 1 is a random intervention group in which half of the patients admitted to the VASLCHCS during study time period will be randomly selected. Providers will see ADE alerts for all patient in the randomly selected experimental group
  Interventions: Behavioral: ADE alert assistant
- Arm 2: Control/No Alerts (No Intervention): The second arm is the control. Alerts will not be displayed for these patients.

INTERVENTIONS:
Behavioral: ADE alert assistant — A note in CPRS alerting providers that patients are at risk for an adverse event based on prescription and lab value histories.
  Arms: Arm 1: ADE Alerts

SUMMARY:
The purpose of this study is to determine if an electronic alerting technology improves time to intervention for possible ADEs, identify what factors affect adoption of ADE alerts, and whether there is a cost benefit associated with the alerting technology.

DETAILED DESCRIPTION:
Inpatient adverse drug events (ADEs) continue to be a major source of morbidity and mortality despite advances in computerized drug safety measures. Reports on the ability of computerized ADE alerts to prevent and mitigate ADEs are lacking. The aims of this project are to 1) Assess organizational, social, and cognitive factors that affect adoption of real-time ADE alerting technology; 2) Analyze the effect of the ADE alerting technology on management and rate of ADEs; and 3) Estimate the cost-benefit of the ADE alerting technology. This study will use a patient randomized design of computerized real-time ADE alerts intended for primary and secondary prevention of ADEs. The ADE alerts promise to reduce mortality, morbidity, and costs due to ADEs. This study will quantify the effect of the alerts in the hands of first-year medical residents and pharmacists. The study will explore the associations of organizational and soci-cognitive barriers and facilitators with the adoption of the ADE alert technology. At the cognitive level, it will explore whether ADE Alerts change user bias in diagnosing ADEs or whether the alerts heighten sensitivity to drug problems.

ELIGIBILITY:
Inclusion Criteria:

- All patients admitted to the SLCVAMC at time of study.

Exclusion Criteria:

- There are no exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R. Nebeker, MD MS, Principal Investigator — VA Health Care Salt Lake City
Locations (1):
- VA Health Care Salt Lake City, Salt Lake City, Utah, United States

REFERENCES:
- [Background] LaFleur J, McAdam-Marx C, Alder SS, Sheng X, Asche CV, Nebeker J, Brixner DI, Silverman SL. Clinical risk factors for fracture among postmenopausal patients at risk for fracture: a historical cohort study using electronic medical record data. J Bone Miner Metab. 2011 Mar;29(2):193-200. doi: 10.1007/s00774-010-0207-y. Epub 2010 Aug 6. PMID 20686803
- [Result] Rupper RW, Bair BD, Sauer BC, Nebeker JR, Shinogle J, Samore M. Out-of-pocket pharmacy expenditures for veterans under medicare part D. Med Care. 2007 Oct;45(10 Supl 2):S77-80. doi: 10.1097/MLR.0b013e3180413871. PMID 17909387
- [Result] Weir CR, Nebeker JR. Critical issues in an electronic documentation system. AMIA Annu Symp Proc. 2007 Oct 11;2007:786-90. PMID 18693944
- [Result] Nebeker JR, Yarnold PR, Soltysik RC, Sauer BC, Sims SA, Samore MH, Rupper RW, Swanson KM, Savitz LA, Shinogle J, Xu W. Developing indicators of inpatient adverse drug events through nonlinear analysis using administrative data. Med Care. 2007 Oct;45(10 Supl 2):S81-8. doi: 10.1097/MLR.0b013e3180616c2c. PMID 17909388
- [Result] Boockvar KS, Livote EE, Goldstein N, Nebeker JR, Siu A, Fried T. Electronic health records and adverse drug events after patient transfer. Qual Saf Health Care. 2010 Oct;19(5):e16. doi: 10.1136/qshc.2009.033050. Epub 2010 Aug 19. PMID 20724395
- [Result] Kaafarani HM, Rosen AK, Nebeker JR, Shimada S, Mull HJ, Rivard PE, Savitz L, Helwig A, Shin MH, Itani KM. Development of trigger tools for surveillance of adverse events in ambulatory surgery. Qual Saf Health Care. 2010 Oct;19(5):425-9. doi: 10.1136/qshc.2008.031591. Epub 2010 May 31. PMID 20513790
- [Result] Olola CH, Rowan B, Narus S, Smith M, Hastings T, Poynton M, Nebeker J, Hales J, Evans RS. Implementation of an emergency medical card and a continuity of care report using continuity of care standard. Methods Inf Med. 2009;48(6):519-30. doi: 10.3414/ME09-01-0003. Epub 2009 Nov 5. PMID 19893849

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: ADE Alerts | Arm 2: Control/No Alerts
Started | 297 | 298
Completed | 297 | 298
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: ADE Alerts | Arm 2: Control/No Alerts | Total
Number analyzed (Participants) | 297 | 298 | 595
Age, Customized [Number; unit: participants]
  18+ | 297 | 298 | 595
Sex/Gender, Customized [Number; unit: participants] — No demographics were collected including gender.
  participants
    Female or Male | NA — No demographics were collected including gender. | NA — No demographics were collected including gender. | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 297 | 298 | 595

OUTCOME MEASURES:

1. Primary Outcome: Time to Intervention Once an ADE Alert Has Fired in CPRS
Time Frame: From the time an ADE alert fires in CPRS until the time action has been taken, i.e. an order placed, up to 24 hours.
Measure: Median (Inter-Quartile Range); unit: hours to intervention
Arm/Group | Arm 1: ADE Alerts | Arm 2: Control/No Alerts
Number analyzed (Participants) | 297 | 298
hours to intervention | 6.8 [1.4 to 25.5] | 8 [1.7 to 42]
Statistical Analysis 1: Comparison: Arm 1: ADE Alerts vs Arm 2: Control/No Alerts; Test type: Superiority or Other; p = 0.6680, Regression, Cox; Cox Proportional Hazard = 0.9396, 95% CI 2-sided [0.7068 to 1.2490]

ADVERSE EVENTS:
Groups:
- Arm 2: Control/No Alert: The second arm is the control. Alerts will not be displayed for these patients.
Arm/Group | Arm 1: ADE Alerts | Arm 2: Control/No Alert
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/298
Other Adverse Events (participants affected / at risk) | 0/297 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes